CLINICAL TRIAL: NCT01288937
Title: A Placebo Controlled, Randomized, Double Blind Trial of Milnacipran for the Treatment of Idiopathic Neuropathy Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Columbia University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Thomas Brannagan, Professor of Clinical Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAF3404
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Idiopathic Peripheral Neuropathy
Keywords: Milnacipran; Idiopathic Peripheral Neuropathy; Diabetic neuropathy; Neuropathic pain
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Milnacipran (Experimental): Patients will receive Milnacipran
  Interventions: Drug: Milnacipran
- Placebo (Placebo Comparator): Patients will receive Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — Patients will be randomly assigned to receive milnacipran 100 mg/day (including a 1 week dose titration period):
  Day 1: 12.5 mg once Day 2, 3: 25 mg/day (12.5 mg twice daily) Day 4, 7: 50 mg/day (25 mg twice daily) After Day 7: 100 mg/day (50 mg twice daily)
  Other Names: Savella
  Arms: Milnacipran
Drug: Placebo — Patients will be randomly assigned to placebo for 9 weeks (including a 1 week dose titration period), matching the schedule of the study drug.
  Other Names: Placebo Pill
  Arms: Placebo

SUMMARY:
This is an 11-week randomized, double-blind, placebo-controlled trial of Milnacipran 100 mg/d in patients with idiopathic neuropathic pain. Milnacipran, a dual norepinephrine and serotonin reuptake inhibitor has been a safe and beneficial treatment for patients with fibromyalgia and may be useful to treat patients with painful peripheral neuropathy.

The primary outcome will be assessed by the change in daily averaged weekly 0-10 pain intensity score, from baseline to week 9, by intention to treat analysis. The same analysis will be used on several secondary measures including daily averaged weekly 0-10 pain intensity score the sleep interference scale and the Rand-36 quality of life scale.

DETAILED DESCRIPTION:
Milnacipran helps serotonin and noradrenaline work more effectively on the central nervous system. Serotonin and noradrenaline are molecules made by the brain that affect how your body responds to pain. Milnacipran, a dual norepinephrine and serotonin reuptake inhibitor has been a safe and beneficial treatment for patients with fibromyalgia and may be useful to treat patients with painful peripheral neuropathy. Many clinical trials for neuropathy pain are done in patients with diabetic neuropathy. Idiopathic neuropathy however, is a common cause of neuropathy and accounts for 25% of all neuropathies, and over 50% of small fiber neuropathies. The information in this study will provide information on whether milnacipran also provide benefit as a medication for neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 to 80 years
* Patients with signs and symptoms of a peripheral neuropathy, with either abnormal nerve conductions or abnormal epidermal nerve fiber density with neuropathic pain.
* Pain will have been present for at least 6 months
* Patients may be on other medications for neuropathic pain (eg, antiepileptic medications, opiates or non steroidal antiinflammatories); however they must be on a stable dose for 4 weeks prior to, with no plan to change during the study
* All patients must have had a normal fasting glucose or B12, thyroid stimulating hormone, and serum protein electrophoresis, since the onset of their symptoms.

Exclusion Criteria:

* Other cause of neuropathy (eg, diabetic neuropathy, toxic neuropathy, HIV neuropathy, celiac neuropathy, inherited neuropathy)
* Unstable angina
* Use of another serotonin and norepinephrine reuptake inhibitors (eg, duloxetine, venlafaxine), tricyclic antidepressants, monoamine oxidase inhibitors (MAOI) or selective serotonin reuptake inhibitors
* Myocardial infarction stroke or life threatening arrhythmia within the last 6 months
* HIV infection
* Hepatic or renal failure
* Pregnancy
* narrow angle glaucoma
* History of epilepsy or a seizure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04-05 (Actual); Primary Completion 2014-10-22 (Actual); Study Completion 2014-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Brannagan III, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be recruited from the practices of the investigators of the peripheral neuropathy center. These subjects will already be receiving treatment in the clinics and private practices of neurologists at the Neurological Institute.
  Patients will also be recruited from physician referrals and advertising.
Pre-assignment Details: Prior to randomization, subjects are assessed at baseline with neurological examinations, physical examination and pain questionnaire/diary.
Groups:
- Placebo: Patients will be randomly assigned to placebo for 9 weeks (including a 1 week dose titration period).
Period: Overall Study
Arm/Group | Milnacipran | Placebo
Started | 4 | 2
Completed | 3 | 2
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milnacipran | Placebo | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Likert Pain Scale Score
Description: The Likert Pain Scale Score is a psychometric scale commonly involved in research that employs questionnaires to measure the intensity of pain. It is used to determine the level of pain for research participants. The minimum score of 0 indicates "no pain" which is the better score and the maximum and total score of 10 indicates the "the worst possible pain" which is the worse outcome . Scores 1-3= Mild, scores 4-6= Moderate, scores 7-10= Severe. It is the most widely used approach to scaling responses in survey research. Patients will fill out a pain diary from baseline to end of treatment. This will be used to assess if there was a reduction in pain of the daily averaged weekly 0-10 pain scale at week 9 compared to the baseline. The Unit of Measure is the scores on the scale.
Time Frame: Baseline, 9 weeks
Population: For the milnacipran arm, 4 subjects were enrolled; however, 1 subject did not complete the study (due to AE: stomach pain) and was not included in the outcome measure data collection/analysis.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 3 | 2
Scores on a scale
  Baseline | 5.6 [3.1 to 8] | 7.15 [5.7 to 8.6]
  9 Weeks | 3.2 [1.4 to 6.6] | 5.15 [4.3 to 6]

ADVERSE EVENTS:
Time Frame: Baseline to 9 weeks.
Description: The definition of adverse event (AE) and/or serious adverse event used to collect AE information is the same as the ClinicalTrials.gov definitions.
Arm/Group | Milnacipran | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 2/4 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=4) | Placebo (N=2)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated and target accrual was unmet due to pre-screening exclusion criteria: 1) excluded concomitant medicines; and 2) patients who had prediabetes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes